CLINICAL TRIAL: NCT00544206
Title: Comparison of Enteral Products for Tube Fed Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Director Clinical Research Operations, Abbott Nutrition
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BK07
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- #1 (Experimental): Diabetes specific enteral feeding product
  Interventions: Other: Diabetes specific feeding product
- #2 (Active Comparator): Standard enteral feeding product
  Interventions: Other: standard enteral feeding product

INTERVENTIONS:
Other: standard enteral feeding product — 16 hrs daily x 5 days
  Arms: #2
Other: Diabetes specific feeding product — 16 hrs daily for 5 days
  Arms: #1

SUMMARY:
To compare the glucose response in tube fed subjects with type 2 diabetes of a standard enteral product to that of a diabetes-specific enteral product

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent
* diagnosis of type 2 diabetes
* HbA1c between 7.0 and 9.0%
* 18 - 75 years of age
* currently receiving a standard enteral product
* anticipated duration on tube feeding at least one month
* 100% of patient's nutrient and energy needs are anticipated to be met by enteral nutrition support
* anticipated life expectancy is more than or equal to 6 months
* free of infections
* no change in medications within 2 weeks prior to screening that could profoundly affect blood glucose

Exclusion Criteria:

* composition of either product is inappropriate for the patient due to allergies or intolerance to any ingredient found in the study products
* composition of either product is inappropriate for the patient due to protein, fluid or electrolyte restrictions for concomitant conditions
* significant cardiovascular event less than or equal to 2 weeks prior to study entry
* major surgery less than or equal to 2 weeks prior to study entry
* pre-planned surgery during the study period
* active malignancy, including melanoma and excluding cutaneous malignancies
* severe dementia
* known allergies to medical grade adhesives and/or skin disinfectants
* taking octreotide
* chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV
* participation in a concomitant trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
mean glucose level | 24 hours

SECONDARY OUTCOMES:
fasting capillary blood glucose level;percentage change from baseline in the dose and amount of antihyperglycemic medication(s), including insulin | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Sacks, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Segal Institute for Clinical Research, Miami, Florida, United States

REFERENCES:
- [Derived] Alish CJ, Garvey WT, Maki KC, Sacks GS, Hustead DS, Hegazi RA, Mustad VA. A diabetes-specific enteral formula improves glycemic variability in patients with type 2 diabetes. Diabetes Technol Ther. 2010 Jun;12(6):419-25. doi: 10.1089/dia.2009.0185. PMID 20470226